CLINICAL TRIAL: NCT01589783
Title: Evaluation of the Influence of Education, Knowledge and Existing Guidelines on the Consumption of Vitamin D During Pregnancy.
Brief Title: Vitamin D During Pregnancy
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: VitDand Preg-HMO-CTIL
Record Dates: First submitted 2012-04-01; First posted 2012-05-02 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Vitamin D Deficiency
Keywords: Pregnancy; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant or newly post partum women
  Interventions: Other: completion of a questionnaire; Other: Blood draw
- family practice physicians and obstetricians
  Interventions: Other: completion of a questionnaire

INTERVENTIONS:
Other: completion of a questionnaire — Completion of a questionnaire
Other: Blood draw — A subset of 100 women will have a blood test to measure Vitamin D levels
  Groups: Pregnant or newly post partum women

SUMMARY:
Vitamin D insufficiency is common globally. Pregnant women, who need an increased supply of this vitamin for the proper development of the fetus, are a significant risk group. The purpose of this study is to examine which factors - education, knowledge from non-professional sources, recommendations from medical staff - influence the use of vitamin D among pregnant women in light of the lack of a clear health policy, and to help formulating guidelines for a new health policy with specific recommendations for vitamin D dosage in pregnancy.

ELIGIBILITY:
Inclusion Criteria for the pregnant of newly post-partum women:

* women between 18-50
* pregnant or just given birth and still hospitalized
* understand and can read Hebrew

Exclusion Criteria:

* those who do not understand or read Hebrew

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We are recruiting either pregnant women or those who just gave birth (and still hospitalized) and a group of both family practice physicians and obstertricians.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Use of Vitamin D in Pregnant Women | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel